CLINICAL TRIAL: NCT03939078
Title: Fractional Ablative CO2 Laser in the Treatment of the Genitourinary Syndrome of Menopause
Brief Title: CO2 Laser in the Treatment of the GSM - (Genitourinary Syndrome of Menopause) Genitourinary Syndrome of Menopause
Status: Completed | Type: Observational
Sponsor: Universidade Federal Fluminense (Other)
Collaborators: Alma Lasers (Industry)
Responsible Party: Principal Investigator, Maria Claudia Almeida Issa, Professor, Universidade Federal Fluminense
Other Study IDs: CO2 laser
Record Dates: First submitted 2019-04-23; First posted 2019-05-06 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Menopause; Vaginal Atrophy; Urinary Incontinence
Keywords: menopause; vaginal atrophy; urinary incontinence; CO2 laser; fractional laser; dyspareunia; vaginal dryness; vaginal lubrication
MeSH Terms: conditions — Urinary Incontinence; Dyspareunia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Vaginal Laser Intervention: Patients will be submitted to vaginal biopsy before and after three laser sections, and therefore will be their own comparative group to see the improvement associated with the laser effects.
  Interventions: Radiation: CO2 fractional ablative laser

INTERVENTIONS:
Radiation: CO2 fractional ablative laser — 3 intravaginal fractional ablative CO2 laser sessions, with one month interval between them.

SUMMARY:
Menopause is a woman's hormonal status one year after her ovulatory failure, when the decrease of circulating estrogen levels leads to a group of symptoms named Genitourinary Syndrome of Menopause (GSM), such as: vaginal dryness, dyspareunia, dysuria, epithelial fragility with recurrent bleedings, loss of genital elasticity and pH alterations causing recurrent infections. The CO2 laser is a fractional ablative source of light, capable of inducing neocollagenesis within the skin, reversing atrophies, increasing blood supply and reorganizing the architectural structure of the treated epithelium. Recent studies in the laser field show great improvement of the SGM, with satisfying results in female's sexual disfunction. Nevertheless, there is still a lack of studies that show, at the same time, the improvement in both patient's subjective reports and objective measurements, such as cytology, histology and immunohistochemistry. This study aims to thoroughly analyze the benefits of the CO2 laser in the treatment of the GMS, comparing the improvement found in questionnaires to the results of cytology, histology and immunohistochemistry for collagen I and III from vaginal biopsies before and after the laser treatment. Therefore, fourteen women after menopause complaining of symptoms of the GSM were selected from the ambulatory of the Hospital Universitário Antônio Pedro. The patients will be submitted to three CO2 intravaginal laser (Femilift®), with a 30-days interval between them. Biopsies of the vaginal wall will be taken one month before the start and one month after the end of the laser sessions, and material will be sent to histology, cytology and immunohistochemistry analysis. Results obtained will be compared to the patients' reports, in order to evaluate subjective and objective improvement due to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women from 40 to 70 years old;
* Post- menopausa (at least one year after cessation of periods);
* Experimenting any symptom related to the Genitourinary Syndrome of Menopause (GSM), such as: vaginal dryness, dyspareunia, urinary incontinence, dysuria, recurrent urinary infections;
* Regular follow up in gynecologist, with recent normal pap smear.

Exclusion Criteria:

* The volunteers must not be under any treatment for this syndrome;
* Volunteers cannot be using hormones or any vaginal treatment;
* Volunteers cannot have previous history of vaginal / uterine cancer;
* Volunteers cannot have previous surgery for urinary incontinence;
* Uterine prolapse;
* Recent altered pap smear.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteer women from 40 to 70 years, healthy and with regular gynecologist follow up, not willing or not eligible to take hormones to treat the GSM, experimenting difficulties in their sexual life and their daily routine, due to vaginal atrophy and urinary incontinence.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Reversion of vaginal atrophy | 1 month after the last (3rd) laser section
  Reversion of vaginal atrophy by the laser stimulation, with increasing layers of epithelial cells, increased collagen deposition and improvement in vascularization.
Improvement in urinary incontinence | 1 month after the third and last laser section
  Improvement in urine involuntary loss, the so called stress incontinence

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Antonio Pedro, Niterói, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] DiBonaventura M, Luo X, Moffatt M, Bushmakin AG, Kumar M, Bobula J. The Association Between Vulvovaginal Atrophy Symptoms and Quality of Life Among Postmenopausal Women in the United States and Western Europe. J Womens Health (Larchmt). 2015 Sep;24(9):713-22. doi: 10.1089/jwh.2014.5177. Epub 2015 Jul 22. PMID 26199981
- [Background] Keil K. Urogenital atrophy: diagnosis, sequelae, and management. Curr Womens Health Rep. 2002 Aug;2(4):305-11. PMID 12150759
- [Background] Palacios S, Castelo-Branco C, Currie H, Mijatovic V, Nappi RE, Simon J, Rees M. Update on management of genitourinary syndrome of menopause: A practical guide. Maturitas. 2015 Nov;82(3):308-13. doi: 10.1016/j.maturitas.2015.07.020. Epub 2015 Jul 26. PMID 26261035
- [Background] Zerbinati N, Serati M, Origoni M, Candiani M, Iannitti T, Salvatore S, Marotta F, Calligaro A. Microscopic and ultrastructural modifications of postmenopausal atrophic vaginal mucosa after fractional carbon dioxide laser treatment. Lasers Med Sci. 2015 Jan;30(1):429-36. doi: 10.1007/s10103-014-1677-2. Epub 2014 Nov 20. PMID 25410301
- [Background] Lindahl SH. Reviewing the options for local estrogen treatment of vaginal atrophy. Int J Womens Health. 2014 Mar 13;6:307-12. doi: 10.2147/IJWH.S52555. eCollection 2014. PMID 24648775
- [Background] Perino A, Calligaro A, Forlani F, Tiberio C, Cucinella G, Svelato A, Saitta S, Calagna G. Vulvo-vaginal atrophy: a new treatment modality using thermo-ablative fractional CO2 laser. Maturitas. 2015 Mar;80(3):296-301. doi: 10.1016/j.maturitas.2014.12.006. Epub 2014 Dec 25. PMID 25596815
- [Background] Hutchinson-Colas J, Segal S. Genitourinary syndrome of menopause and the use of laser therapy. Maturitas. 2015 Dec;82(4):342-5. doi: 10.1016/j.maturitas.2015.08.001. Epub 2015 Aug 12. PMID 26323234
- [Derived] Bretas TLB, Issa MCA, Fialho SCAV, Villar EAG, Velarde LGC, Perez-Lopez FR. Vaginal collagen I and III changes after carbon dioxide laser application in postmenopausal women with the genitourinary syndrome: a pilot study. Climacteric. 2022 Apr;25(2):186-194. doi: 10.1080/13697137.2021.1941850. Epub 2021 Jul 22. PMID 34291703